CLINICAL TRIAL: NCT05871567
Title: Assessment of the DNA Mismatch Repair System is Crucial in Colorectal Cancers Necessitating Adjuvant Treatment: a Propensity Score-matched and Win Ratio Analysis
Brief Title: Predictive Value of DNA Mismatch Repair System in Colorectal Cancers
Acronym: DNAMMR
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Gennaro Galizia, Full Professor of Surgery, University of Campania Luigi Vanvitelli
Other Study IDs: Università Vanvitelli Napoli
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: MSI-H Colorectal Cancer
Keywords: Colorectal cancers;; DNA mismatch repair;; Win ratio
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — specimens from surgical resection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1 or MSS: colorectal cancers (CRCs) with stable microsatellite
  Interventions: Procedure: colorectal resection
- group 2 or MSI: colorectal cancers (CRCs) with unstable microsatellite
  Interventions: Procedure: colorectal resection

INTERVENTIONS:
Procedure: colorectal resection — potential resective surgery

SUMMARY:
* Microsatellite instable (MSI) tumors represent almost the 15% of all sporadic colorectal cancers (CRCs).
* Literature data show that this unique tumor population appears to be poorly responsive to conventional chemotherapy and conversely reveals excellent results to immunotherapy.
* Our data, as demonstrated by propensity score-matched and win ratio analysis, show that there are no substantial differences between MSI and MSS tumors in early CRC stages treated with surgery alone.
* On the contrary, stable tumors (MSS) did much better than MSI tumors in advanced CRC stages undergoing conventional adjuvant treatment.
* Determination of status of DNA mismatch repair system is crucial in high-risk CRCs to optimize treatment.

DETAILED DESCRIPTION:
Colorectal cancers (CRCs) with deficient DNA mismatch repair (MMR) system (so called dMMR or MSI tumors) represent a no-negligible part of sporadic CRCs. Prognostic value of this unique cell population remains controversial, but undoubtedly these tumors are characterized by poor response to conventional chemotherapy, an high tumor mutational burden resulting in a brisk immuno response, and, as recently observed, excellent results to the immunotherapy. The aim of this study was to evaluate, by using sophisticated statistical analyses, the predictive value of MSI status and its optimal treatment.

A series of 403 consecutive CRC patients treated by the same oncological team from 2014 to 2021 entered the study. No patients underwent immunotherapy. Immunohistochemistry, integrated by polymerase chain reaction if appropriate, was used to categorize specimens in microsatellite stable (MSS) and instable (MSI) tumors. The win ratio (WR) approach was utilized to compare composite outcomes of MSS and MSI tumors while controlling for radical versus no radical resection, propensity score-matched analysis, and reversing primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive CRC patients observed from January 2014 to December 2021

Exclusion Criteria:

* Patients with suspected or confirmed Lynch's syndrome (12 patients) and rectal cancers (98 patients) undergoing neoadjuvant treatment

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CRC patients undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
survival rate | "From date of surgical operation until the date of death from any cause assessed up to 60 months"
  overall survival

SECONDARY OUTCOMES:
recurrence rate | "From date of surgical operation until the date of documented tumor recurrence assessed up to 60 months"
  disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Galizia, MD, Study Director — University of Campania 'Luigi Vanvitelli'

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available by contacting the principal investigator
Time Frame: data will become available after conclusion of the trial and publication of the results. After that data will be available for two years.
Access Criteria: gennaro.galizia@unicampania.it